CLINICAL TRIAL: NCT02687347
Title: A Double Blind Randomized Clinical Trial to Investigate the Efficacy and Safety of Ultra-low Dose Methadone as Adjuvant Analgesic Therapy in Cancer Patients With Pain
Brief Title: Efficacy and Safety of Ultra-low Dose Methadone as Adjuvant Analgesic in Cancer Patients With Pain
Acronym: UDOME
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Jordi Perez, Codirector Cancer Pain Program. McGill University Health Centre. Montreal, Canada, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 15-369 MP-CUSM
Record Dates: First submitted 2016-02-08; First posted 2016-02-22 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Pain, Intractable
MeSH Terms: conditions — Pain, Intractable | interventions — Methadone; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- study arm (Experimental): low dose methadone (1-10mg daily)
  Interventions: Drug: oral methadone
- control arm (Active Comparator): low dose morphine (1-10 mg/day)
  Interventions: Drug: oral morphine

INTERVENTIONS:
Drug: oral methadone — Oral methadone is the study drug
  Arms: study arm
Drug: oral morphine — Oral morphine is the active comparator. It is not a placebo intervention
  Arms: control arm

SUMMARY:
The research hypothesis of this study is: In patients with moderate to severe cancer related pain, the addition of low dose methadone to an existing opioid significantly reduces pain severity compared to low doses morphine.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed of cancer-related pain of more than 3 months duration
* Pain relief during the last week rated unsatisfactory by the patient
* Pain severity during the last week rated moderate (between 4 and 7/10)
* Analgesic therapy must have been stable for 7 days
* Able to understand English or French
* Willing and able to give written informed consent

Exclusion Criteria:

* Patients who are currently receiving or have received methadone as analgesic in the last 6 months
* Contraindication to receive methadone (allergy, QTc segment on the ECG>450msec, concurrent treatment with medication that could increase methadone's effects)
* Patients presenting with changes in their cancer status/treatment with potential effects on their pain severity, during the duration of the trial (eg: new metastasis, indication for radiotherapy)
* Patients whose life expectancy is shorter than 2 months
* Patients with cognitive impairment presenting with difficulties understanding the trial and completing the research questionnaires
* Pregnant or lactating women (women of childbearing potential must have negative pregnancy test)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2016-02; Primary Completion 2018-02 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
pain relief | 2 months
  1) Pain item of the Edmonton Symptom Assessment Scale
pain relief | 2 months
  Questions 3 to 6 of the Brief Pain Inventory

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0". | 2 months
  prevalence and severity of opioid induced side effects

OTHER OUTCOMES:
pain interference | 2 months
  Brief Pain Inventory: Composite questions 9-A to 9-G

CONTACTS AND LOCATIONS:
Locations (1):
- Alan Edwards Pain Management Unit. Mcgill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
1. Demographic, cancer status, pain medication, symptom severity and side effects profile will be collected for each participant throughout the study
  2. Data will be collected by clinical interview with research nurse
  3. Data will be available to researchers immediately